CLINICAL TRIAL: NCT02507284
Title: An Exploratory Phase II Study to Determine the Tolerability, Safety, and Activity of a Novel Vasopressin 1a Receptor Antagonist (SRX246) in Irritable Subjects With Huntington's Disease (HD)
Brief Title: Tolerability, Safety, and Activity of SRX246 in Irritable Subjects With Huntington's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azevan Pharmaceuticals (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); NeuroNEXT Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVN011; 1U44NS090616-01A1 (NIH)
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Irritable Mood; Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — SRX246

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SRX246 120mg BID (Experimental): SRX246 capsules, administered orally, in divided doses twice daily
  Interventions: Drug: SRX246
- SRX246 160mg BID (Experimental): SRX246 capsules, administered orally, in divided doses twice daily
  Interventions: Drug: SRX246
- Placebo (Placebo Comparator): Placebo capsules, administered orally, in divided doses twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRX246
  Arms: SRX246 120mg BID; SRX246 160mg BID
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the tolerability, safety and activity of SRX246 in the treatment of irritability in patients with Huntington's disease. Two-thirds of all participants will receive SRX246, while the other third will receive a placebo.

DETAILED DESCRIPTION:
SRX246 is a first-in-class vasopressin 1a (V1a) receptor antagonist that crosses the blood-brain barrier following oral administration. The molecule exhibits high affinity and high selectivity for its target receptor. Preclinical pharmacology studies have demonstrated significant CNS effects in models of irritability, including impulsive aggression, depression, and anxiety. In an experimental medicine fMRI study in healthy volunteers, SRX246 treatment significantly attenuated the effect of intranasal AVP in brain circuits known to modulate emotional responses to stimuli that elicit aggression/fear. Together, these findings suggest that SRX246 has potential as a novel therapeutic agent for major neuropsychiatric symptoms seen in HD patients.

This is a 3-arm, multicenter, randomized, placebo-controlled, double-blind, 12 week, dose escalation study of SRX246 in irritable Subjects with early symptomatic HD.

Following an initial screening visit, Subjects fulfilling the study inclusion and exclusion criteria will enter a pre-treatment screening phase to permit evaluations to confirm eligibility for inclusion into the study. This screening phase will be no longer than 30 days. At the completion of the screening period, eligible Subjects will be randomized at baseline visit to receive either placebo or final doses of SRX246 of 120 mg twice daily or 160 mg twice daily during the double-blind treatment phase. At baseline, Subjects in the active groups will receive 80 mg twice daily for 2 weeks, then escalate to 120 mg twice daily for 4 weeks. Then one group of Subjects will continue to take 120 mg of SRX246 twice daily for an additional 6 weeks, and the second group of Subjects will increase their dose to 160 mg of SRX246 twice daily for 6 weeks. Total dosing duration is 12 weeks.

Subjects in the placebo group will receive a similar number of capsules that are identical in appearance to the capsules that contain SRX246 during the trial, in order to preserve the blind.

In all groups, dose escalation will occur (stepwise) if patients have not experienced dose-limiting adverse effects. Patients who cannot tolerate their final dose of drug (or placebo) can have this dose reduced without compromising the blinding.

Subjects will have periodic visits either "in-person" or by "telephone", to assess tolerability, safety, and several measures of irritability and other problem behaviors, and clinical assessments for activity signals.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female Subjects aged 18 years or older
2. Subjects must have clinical features of HD, which can include motor, cognitive, or behavioral symptoms
3. A confirmatory family history of HD; OR CAG repeat expansion ≥ 37
4. Total Functional Capacity (TFC) score of 5-13
5. Evidence of irritability; a score of at least 2 or greater on the severity measure of either the UHDRS Irritability question (30b) or Aggression question (Disruptive or Aggressive Behavior, 31b)
6. Women of childbearing potential (i.e., those not postmenopausal or surgically sterile) must have a negative pregnancy test, be non-lactating and use adequate contraception methods during the study. Adequate birth control includes: abstinence; oral, implanted or injected contraceptives, e.g., birth control pills; intra-uterine device; barrier (vaginal ring or diaphragm/cervical cap with spermicide); transdermal patch. Reliable contraception must have been in use 30 days prior to the Baseline Visit. Partner(s) contraception (e.g., male partner with vasectomy or other surgical contraception) is acceptable.
7. Men must agree not to father a child during the study and one month after and to use contraception. Barrier with spermicide or surgical contraception is acceptable. Partner(s) contraception (e.g., female partner taking birth control pills or surgically sterile) is acceptable.
8. Subjects must be able to swallow study drug capsules whole.
9. Sufficient English skills to complete all assessments without assistance of an English language interpreter. Subjects with HD who cannot read or write might qualify for enrollment in the study. Site PIs will have to decide in each case whether the Subject can understand and fully participate with help from his/her Informant.
10. Availability of a responsible Informant (referred to as a "study partner" in the consent document) who has good English skills, is familiar with the Subject, and is able and willing to comply with all required study procedures, ensuring that the patient attends all study visits and takes the study medicine as instructed. The study partner must spend time with the patient a minimum of 4 times per week on 4 separate days, and must monitor the patient's compliance and adverse events, participate in caregiver assessments, and use the eDiary.
11. Subject has provided written, informed consent or, if Subject lacks the capacity to provide informed consent (as determined by an independent assessment by a qualified healthcare provider not directly involved in other study activities), a legally authorized representative (LAR) has provided written informed consent and the Subject has provided assent.

Exclusion Criteria:

1. Any significant neurologic disease other than HD at Screening.
2. Severe psychotic features or other severe psychiatric symptoms within the last three months which could lead to difficulty complying with the protocol.
3. History of active alcohol or substance abuse within the past two years or Subject is unable to refrain from substance abuse throughout the study.
4. Any chronic disability, significant systemic illness or unstable medical condition at Screening or Baseline that could lead to difficulty complying with the protocol.
5. Use of any investigational drugs within 30 days of Screening.
6. Subject has known allergy to any of the components of study medication.
7. Subject is currently pregnant, breast-feeding and/or lactating.
8. Subject acknowledges present use of illicit drugs at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - University of Alabama, Birmingham, Alabama
  - UCLA, Neurology Clinic, Los Angeles, California
  - UC Davis Medical Center, Department of Neurology, CTSC Clinical Research Center, Sacramento, California
  - University of Colorado Hospital Translational Research Center, Aurora, Colorado
  - University of Miami, Miller School of Medicine, Jackson Behavioral Health Hospital, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Out-Patient Neurology Clinic, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Stony Brook Clinical Research Center, Department of Neurology, East Setauket, New York
  - Columbia University Medical Center, New York Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University Medical Arts Building, Cincinnati, Ohio
  - Ohio State University, Wexner Medical Center, Department of Neurology, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Department of Neurology, Pittsburgh, Pennsylvania
  - Vanderbilt Clinical Research Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah, Department of Neurology, Salt Lake City, Utah
  - University of Virginia Health System, Department of Neurology, Charlottesville, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- SRX246 120mg BID; SRX246 160mg BID: SRX246 capsules, administered orally, in divided doses twice daily
  SRX246
- Placebo: Placebo capsules, administered orally, in divided doses twice daily
  Placebo
Period: Overall Study
Arm/Group | SRX246 120mg BID | SRX246 160mg BID | Placebo
Started | 36 | 34 | 36
Completed | 25 | 27 | 30
Not Completed | 11 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SRX246 120mg BID | SRX246 160mg BID | Placebo | Total
Number analyzed (Participants) | 36 | 34 | 36 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (13.2) | 48.9 (12.7) | 51.7 (10.4) | 50.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 20 | 55
  Male | 18 | 17 | 16 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36 | 33 | 36 | 105
  Not White | 0 | 1 | 0 | 1
  Hispanic/Latino | 2 | 4 | 0 | 6
  Not Hispanic/Latino | 34 | 30 | 35 | 99
  Missing | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 36 | 34 | 36 | 106

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of SRX246
Description: The primary endpoint, tolerability of SRX246, was assessed by the number of completers in each group.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SRX246 120mg BID | SRX246 160mg BID | Placebo
Number analyzed (Participants) | 36 | 34 | 36
Participants | 25 | 27 | 30

2. Secondary Outcome: Safety of SRX246
Description: The Safety of SRX246 was assessed by the number of participants who experience an adverse event.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SRX246 120mg BID | SRX246 160mg BID | Placebo
Number analyzed (Participants) | 36 | 34 | 36
Participants | 29 | 30 | 26
Statistical Analysis 1: Comparison: SRX246 120mg BID vs SRX246 160mg BID vs Placebo; Test type: Non-Inferiority — Results for the secondary safety endpoint, adverse events (AEs) in study subjects, was performed using a test for non-inferiority with a threshold of 0.50. The null hypothesis is that the treatment minus placebo proportion difference is greater than (or equal to) the margin of 0.50 and the alternative hypothesis is that the difference is less than 0.50; p = 0.50, t-test, 1 sided; Risk Ratio (RR) = 0.025

ADVERSE EVENTS:
Time Frame: From first dose of study drug to last date of patient follow-up at end of study (an average of 12-weeks)
Description: The data are reported based on 3 arms: SRX246 120mg, SRX246 160mg and Placebo. All subjects were randomized at the beginning of the study to one of those 3 arms. Thus, the data are displayed this way, even though all participants randomized to the SRX246 arms received a starting dose of SRX246 80mg, then escalated to SRX246 120mg, and then the group that was randomized to the SRX246 160mg was dose escalated.
Groups:
- SRX246 120mg BID: SRX246 capsules, administered orally, in divided doses twice daily. This group includes those participants that were enrolled and randomized to the group assigned to receive 120mg BID throughout the study. The data are reported based on 3 arms: SRX246 120mg, SRX246 160mg and Placebo. All subjects were randomized at the beginning of the study to one of these 3 arms. Thus, the data are displayed this way, even though all participants randomized to the SRX246 arms received a starting dose of SRX246 80mg, then escalated to SRX246 120mg, and then the group that was randomized to the SRX246 160mg was dose escalated.
- SRX246 160mg BID: SRX246 capsules, administered orally, in divided doses twice daily. This group includes those participants that were enrolled and randomized to the group assigned to receive 160mg BID throughout the study. The data are reported based on 3 arms: SRX246 120mg, SRX246 160mg and Placebo. All subjects were randomized at the beginning of the study to one of those 3 arms. Thus, the data are displayed this way, even though all participants randomized to the SRX246 arms received a starting dose of SRX246 80mg, then escalated to SRX246 120mg, and then the group that was randomized to the SRX246 160mg was dose escalated.
Arm/Group | SRX246 120mg BID | SRX246 160mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 5/36 | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 29/36 | 30/34 | 26/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SRX246 120mg BID (N=36) | SRX246 160mg BID (N=34) | Placebo (N=36)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aggression and Irritability (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SRX246 120mg BID (N=36) | SRX246 160mg BID (N=34) | Placebo (N=36)
nausea (Gastrointestinal disorders) | 7 (13) | 9 (13) | 4 (4) — Including gastrointestinal upset, vomiting, abdominal pain, dyspepsia
Fatigue (General disorders) | 3 (3) | 5 (7) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (7) | 4 (4) | 9 (11) — including urinary tract infection
Fall (Injury, poisoning and procedural complications) | 4 (6) | 4 (7) | 5 (5) — including ankle fracture, contusion
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (6) | 1 (1)
headache (Nervous system disorders) | 6 (7) | 4 (6) | 8 (9) — including lethargy, dizziness, paraesthesia
depressed mood (Psychiatric disorders) | 8 (11) | 8 (9) | 4 (6) — including insomnia, irritability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT02507284/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT02507284/SAP_001.pdf